CLINICAL TRIAL: NCT06472830
Title: Monoclonal Gammopathy of Undetermined Significance (MGUS) /Myeloma Awareness and Genetic Insights Campaign (MAGIC) Screening Study
Brief Title: Prevalence of Monoclonal Gammopathy of Undetermined Significance (MGUS) / Multiple Myeloma (MM) Among Unique Populations of Black People
Acronym: MAGIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-008956; NCI-2024-04825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008956 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants undergo medical chart review and blood sample collection, as well as complete a questionnaire on study. Participants who test positive for MGUS are notified, along with their primary care physician, so that the necessary follow up and referral is provided as clinically indicated.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to screen for monoclonal gammopathies in people of East African descent. Monoclonal gammopathy is a condition where abnormal proteins are found in the blood, most commonly called monoclonal gammopathy of undetermined significance or MGUS. There is little information on the presence of this condition in people of East African descent. This study is being done to determine how this condition affects this population in order to better treat and/or prevent this condition in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the prevalence of monoclonal gammopathies (MGUS, Smoldering and Multiple Myeloma) in people of East African descent in Minnesota.

OUTLINE: This is an observational study.

Participants undergo medical chart review and blood sample collection, as well as complete a questionnaire on study. Participants who test positive for MGUS are notified, along with their primary care physician, so that the necessary follow up and referral is provided as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 40 years
* Self-reported east African ancestry (including individuals of mixed east African descent)
* Willing and able to review, understand, and provide consent before starting any study-specific procedures

Exclusion Criteria:

* Pregnant women

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who self-report east African ancestry without a diagnosis of multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of MGUS in people of east African descent | Up to 10 years
  Screening for MGUS using mass spectrometry to detect monoclonal proteins among people of east African descent in Minnesota.

CONTACTS AND LOCATIONS:
Overall Officials: Joselle M. Cook, M.B.B.S., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials